CLINICAL TRIAL: NCT03634293
Title: PCSK9 Inhibitor: a New Tool to Fight Septic Shock
Brief Title: Treatment of Severe Infection With Antihyperlipidemia Drug
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wolfson Medical Center (Other Government)
Collaborators: Assaf-Harofeh Medical Center (Other Government); Sanofi (Industry)
Responsible Party: Principal Investigator, Rozman Ziv, Principal investigator, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PCSK9 administration in sepsis
Record Dates: First submitted 2018-07-30; First posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Sepsis; Septic Shock
Keywords: sepsis; septic shock; PCSK9 INHIBITOR
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — alirocumab; Saline Solution

STUDY DESIGN:
Intervention Model Description: the study is a randomized placebo controlled double blinded study. the control group will be receiving placebo and the treatment group will be receiving the study drug.
Who Masked: Participant, Care Provider, Investigator
Masking Description: the study drug and placebo will be identical arriving from the manufacturing company as a clear fluid for subcutaneous injection of 2 ml'. both arms, the control and intervention, will receive identical subcutaneous injections. the randomization will be prior to recruitment in the pharmacy. At the end of the study the outcomes assessor will be exposed to the data unblended.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Placebo Comparator): The group will receive 2 ml' saline subcutaneous injection upon randomization when admitted to the ICU with the diagnosis of sepsis or septic shock
  Interventions: Drug: Saline Solution
- treatment group (Active Comparator): The group will receive a 2 ml' subcutaneous injection of the study drug Alirocumab 150 mg', upon randomization when admitted to the ICU with the diagnosis of sepsis or septic shock.
  Interventions: Drug: Alirocumab Injectable Product

INTERVENTIONS:
Drug: Alirocumab Injectable Product — Alirocumab is an human monoclonal antibodies directed against Proprotein convertase subtilisin/kexin type 9 (PCSK9). It is administered once every two weeks subcutaneously.
  Other Names: Praluent
  Arms: treatment group
Drug: Saline Solution — The placebo will be 2 ml' of 0.9% saline injected subcutaneously.
  Arms: control group

SUMMARY:
Proprotein convertase subtilisin kexin 9 (PCSK9) inhibitors increase LDL receptors by decreasing its degradation. In sepsis the pathogenic substances, endotoxin, lipoteichoic acid, phospholipomannan are the main cause of the ongoing inflammation that causes the severe damage and outcome. these substances are removed from the blood by the LDL receptors. By administering PCSK9 inhibitors to patients with sepsis/septic shock this inflammatory response can be stopped and by doing so improve the patients outcome.

DETAILED DESCRIPTION:
Sepsis is a life-threatening organ dysfunction caused by a dysregulated host response to infection with a high mortality rate. The main causative agents in the ICU to cause sepsis and septic shock are gram negative bacteria Klebsiella spp., Escherichia coli (E. coli), and Pseudomonas aeruginosa (P. aeruginosa) and gram positive Staphylococcus aureus (S. aureus), Streptococcus pyogenes (S. pyogenes). The role of bacterial endotoxin is known to be central to development of septic shock in gram-negative bacterial sepsis. Gram negative bacteria's membranes are made of lipopolysaccharides (LPS), the endotoxin. The pattern recognition receptor for LPS is Toll-like receptor 4 (TLR4), upon activation initiates the inflammatory cascade.

In past studies it was demonstrated that despite the lack of LPS on gram positive bacteria, TLR4 mutant's mice had higher bacterial burden and lower survivability suggesting a role in the inflammatory cascade of TLR4 despite the lack of LPS.

Super antigen bind directly to the major histocompatibility complex II (MHC-II) receptor and T cell receptor causing a massive T cell activation bypassing the antigen presenting cell leading to cytokine storm.

Studies on murine, measuring the levels of LDL during inflammation, demonstrated a high level of LDL in the blood due to suppression of LDL receptor proteins in the liver. Proprotein convertase subtilisin kexin 9 (PCSK9) is a serine protease secreted by the liver binding to the LDL receptor and enhancing its degradation causing the increase of LDL levels in the blood. In the absence of PCSK9, the number of LDL receptors on the liver cell surface increases and more circulating LDL is removed from the plasma.

PCSK9 is found to increase during inflammation. Grefhorst A et al, demonstrated that administration of recombinant PCSK9 to mice reduced hepatic LDL receptors. Based on that finding, Kenneth R. Feingold et al, conducted a study administering lipopolysaccharides (LPS) to mice intra peritoneal, measuring the levels of hepatic LDL receptor protein levels, and PCSK9 messenger ribonucleic acid (mRNA) levels in the liver and in the kidneys. There was an increase in the PCSK9 levels within 4 hours in response to LPS and in response to several other mechanisms causing systemic inflammation.

Microbial pathogenic lipids, namely LPS in gram negative bacteria, lipoteichoic acid in gram-positive bacteria, and phospholipomannan in fungi, are bound to lipids in the blood, causing an increase in PCSK9 in plasma. This led to the speculation that increased lipid clearance by the liver leads to increased LPS clearance affecting the process of sepsis and septic shock. Thus administering PCSK9 inhibitor leading to increase in lipids uptake by the liver would positively affect the septic patient.

The benefit of inhibiting PCSK9 in sepsis is further strengthened by a study of Keith R et al examining septic patients who had at least one PCSK9 loss of function allele that showed increased survival over a 28-day period compared to those with gain of function allele.

A study made by, Berger J M et al, on murines showed lack of benefit in septic mice when administering PCSK9 inhibitor adjacent to LPS injection peritoneally. In this study PCSK9 inhibitor was administered as a monotherapy while in studies showing benefit, antibiotics treatment was given. Furthermore the lack of benefit can be explained by the short duration between the induction of endotoxemia to PCSK9 inhibitors administration, inhibiting the binding of the inflammatory mediators to the lipid transports in the blood prior to the activation of the inflammatory response which is needed. As previously mentioned PCSK9 levels that were measured in past studies only increased after 4 hours from inflammatory induction and not immediately after the exposure to LPS.

Due to the results of studies supporting the clinical benefit of PCSK9 inhibitors the investigators intend to conduct a study in septic patients and septic shock patients upon admission to the ICU.

The PCSK9 inhibitor is a relatively safe drug with a small amount of mild adverse events. In the "ODYSSEY LONG TERM" study with 2341 patients, examining among others the safety of the PCSK9 inhibitor use, Alirocumab, at a dose of 150 mg had similar rates of adverse events between the treatment group and the placebo. The Alirocumab patients had higher rates than the placebo group with injection-site reactions, myalgia, neurocognitive events (amnesia, memory impairment, and confusional state), and ophthalmologic events at low rates. In a recent large meta-analysis examining adverse effects showed no statistical significant regarding neurocognitive events or diabetes. Same results were received in a small post marketing study finding most adverse events of flu like symptoms and myalgia without difference between placebo, Alirocumab 75 mg dose and the 150 mg dose.

In order to validate the clinical use of PCSK9 inhibitor the investigators plan to administer 150 mg subcutaneous injection of Alirocumab upon admission to the ICU to patients diagnosed with sepsis or septic shock every two weeks. Two centers will be participating in the study from Israel.

ELIGIBILITY:
* Inclusion Criteria:

  * Subject is admitted to the ICU
  * Subject has a clinical diagnosis of sepsis or septic shock
* Exclusion Criteria:

  * Liver function tests (aspartate aminotransferase and Alanine transaminase) above three times the normal levels.
  * Creatinine clearance levels below 30.
  * Life expectancy below 28 days due to terminal illness.
  * Moribund condition with life expectancy of less than 24 hours.
  * Pregnancy or lactating women.
  * Known hypersensitivity to the study drug.
  * Grade IV peripheral edema at time of randomization.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 712 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
survival | At 28 days from randomization
  We will measure the survival at 28 days

SECONDARY OUTCOMES:
Length of stay in the ICU | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 month
  Time until discharge from the ICU to the regular wards
Time on vasopressors | From the date of documented use of vasopressor drugs until the documented cessation of this therapy assessed up to 24 month
  The time the patient requires the supports of vasopressors drugs, mainly Norepinephrine
Time on mechanical ventilation | From the date of documented use of mechanical ventilation until the documented discontinuation of mechanical ventilation assessed up to 24 month
  The time the patient requires the support of mechanical ventilation
Levels of inflammatory mediators | At the time of randomization once every day assessed up to 28 days
  The levels of C reactive protein and leukocytes during a time frame
Lactate levels | At the time of randomization and 3 times a day until the documentation of normal lactate values assessed up to 28 days
  The time it takes for lactate levels to return to normal
Length of hospital stay | From the time of randomization until first documentation of hospital discharge or date of death from any cause assessed up to 24 month
  The time the patient is hospitalized in the ICU and the wards

CONTACTS AND LOCATIONS:
Overall Officials: Ziv Rosman, MD, Study Director — Wolfson Medical Center
Locations (1):
- Eduard Ilgiyaev, Rishon LeZiyyon, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Due to the inability to obtain a written consent from the patients at the time of randomization and recruitment, the release of the data will be decided later on with a Helsinki Committee for Human Rights

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Sriskandan S, Cohen J. Gram-positive sepsis. Mechanisms and differences from gram-negative sepsis. Infect Dis Clin North Am. 1999 Jun;13(2):397-412. doi: 10.1016/s0891-5520(05)70082-9. PMID 10340174
- [Background] Medzhitov R, Preston-Hurlburt P, Janeway CA Jr. A human homologue of the Drosophila Toll protein signals activation of adaptive immunity. Nature. 1997 Jul 24;388(6640):394-7. doi: 10.1038/41131. PMID 9237759
- [Background] Ramachandran G. Gram-positive and gram-negative bacterial toxins in sepsis: a brief review. Virulence. 2014 Jan 1;5(1):213-8. doi: 10.4161/viru.27024. Epub 2013 Nov 5. PMID 24193365
- [Background] Branger J, Knapp S, Weijer S, Leemans JC, Pater JM, Speelman P, Florquin S, van der Poll T. Role of Toll-like receptor 4 in gram-positive and gram-negative pneumonia in mice. Infect Immun. 2004 Feb;72(2):788-94. doi: 10.1128/IAI.72.2.788-794.2004. PMID 14742522
- [Background] Liao W, Rudling M, Angelin B. Endotoxin suppresses rat hepatic low-density lipoprotein receptor expression. Biochem J. 1996 Feb 1;313 ( Pt 3)(Pt 3):873-8. doi: 10.1042/bj3130873. PMID 8611169
- [Background] Horton JD, Cohen JC, Hobbs HH. Molecular biology of PCSK9: its role in LDL metabolism. Trends Biochem Sci. 2007 Feb;32(2):71-7. doi: 10.1016/j.tibs.2006.12.008. Epub 2007 Jan 9. PMID 17215125
- [Background] Seidah NG, Awan Z, Chretien M, Mbikay M. PCSK9: a key modulator of cardiovascular health. Circ Res. 2014 Mar 14;114(6):1022-36. doi: 10.1161/CIRCRESAHA.114.301621. PMID 24625727
- [Background] Gouni-Berthold I, Descamps OS, Fraass U, Hartfield E, Allcott K, Dent R, Marz W. Systematic review of published Phase 3 data on anti-PCSK9 monoclonal antibodies in patients with hypercholesterolaemia. Br J Clin Pharmacol. 2016 Dec;82(6):1412-1443. doi: 10.1111/bcp.13066. Epub 2016 Oct 4. PMID 27478094
- [Background] Feingold KR, Moser AH, Shigenaga JK, Patzek SM, Grunfeld C. Inflammation stimulates the expression of PCSK9. Biochem Biophys Res Commun. 2008 Sep 19;374(2):341-4. doi: 10.1016/j.bbrc.2008.07.023. Epub 2008 Jul 16. PMID 18638454
- [Background] Grefhorst A, McNutt MC, Lagace TA, Horton JD. Plasma PCSK9 preferentially reduces liver LDL receptors in mice. J Lipid Res. 2008 Jun;49(6):1303-11. doi: 10.1194/jlr.M800027-JLR200. Epub 2008 Mar 19. PMID 18354138
- [Background] dos Santos C, Marshall JC. Bridging lipid metabolism and innate host defense. Sci Transl Med. 2014 Oct 15;6(258):258fs41. doi: 10.1126/scitranslmed.3010501. PMID 25320231
- [Background] Norata GD, Tavori H, Pirillo A, Fazio S, Catapano AL. Biology of proprotein convertase subtilisin kexin 9: beyond low-density lipoprotein cholesterol lowering. Cardiovasc Res. 2016 Oct;112(1):429-42. doi: 10.1093/cvr/cvw194. Epub 2016 Aug 5. PMID 27496869
- [Background] Walley KR, Francis GA, Opal SM, Stein EA, Russell JA, Boyd JH. The Central Role of Proprotein Convertase Subtilisin/Kexin Type 9 in Septic Pathogen Lipid Transport and Clearance. Am J Respir Crit Care Med. 2015 Dec 1;192(11):1275-86. doi: 10.1164/rccm.201505-0876CI. PMID 26252194
- [Background] Walley KR, Thain KR, Russell JA, Reilly MP, Meyer NJ, Ferguson JF, Christie JD, Nakada TA, Fjell CD, Thair SA, Cirstea MS, Boyd JH. PCSK9 is a critical regulator of the innate immune response and septic shock outcome. Sci Transl Med. 2014 Oct 15;6(258):258ra143. doi: 10.1126/scitranslmed.3008782. PMID 25320235
- [Background] Berger JM, Loza Valdes A, Gromada J, Anderson N, Horton JD. Inhibition of PCSK9 does not improve lipopolysaccharide-induced mortality in mice. J Lipid Res. 2017 Aug;58(8):1661-1669. doi: 10.1194/jlr.M076844. Epub 2017 Jun 9. PMID 28600283
- [Background] Robinson JG, Farnier M, Krempf M, Bergeron J, Luc G, Averna M, Stroes ES, Langslet G, Raal FJ, El Shahawy M, Koren MJ, Lepor NE, Lorenzato C, Pordy R, Chaudhari U, Kastelein JJ; ODYSSEY LONG TERM Investigators. Efficacy and safety of alirocumab in reducing lipids and cardiovascular events. N Engl J Med. 2015 Apr 16;372(16):1489-99. doi: 10.1056/NEJMoa1501031. Epub 2015 Mar 15. PMID 25773378
- [Background] Karatasakis A, Danek BA, Karacsonyi J, Rangan BV, Roesle MK, Knickelbine T, Miedema MD, Khalili H, Ahmad Z, Abdullah S, Banerjee S, Brilakis ES. Effect of PCSK9 Inhibitors on Clinical Outcomes in Patients With Hypercholesterolemia: A Meta-Analysis of 35 Randomized Controlled Trials. J Am Heart Assoc. 2017 Dec 9;6(12):e006910. doi: 10.1161/JAHA.117.006910. PMID 29223954
- [Background] Choi J, Khan AM, Jarmin M, Goldenberg N, Glueck CJ, Wang P. Efficacy and safety of proprotein convertase subtilisin-kexin type 9 (PCSK9) inhibitors, alirocumab and evolocumab, a post-commercialization study. Lipids Health Dis. 2017 Jul 24;16(1):141. doi: 10.1186/s12944-017-0493-7. PMID 28738813
- [Background] Sabatine MS, Giugliano RP, Keech AC, Honarpour N, Wiviott SD, Murphy SA, Kuder JF, Wang H, Liu T, Wasserman SM, Sever PS, Pedersen TR; FOURIER Steering Committee and Investigators. Evolocumab and Clinical Outcomes in Patients with Cardiovascular Disease. N Engl J Med. 2017 May 4;376(18):1713-1722. doi: 10.1056/NEJMoa1615664. Epub 2017 Mar 17. PMID 28304224